CLINICAL TRIAL: NCT00131066
Title: Long-Term Safety Follow-Up Study of Psoriasis Patients Who Have Received MEDI-507
Brief Title: Long-Term Follow-Up Study of Psoriasis Patients
Status: Completed | Type: Observational
Sponsor: MedImmune LLC (Industry)
Responsible Party: Barbara White, MedImmune Inc.
Other Study IDs: MI-CP085
Record Dates: First submitted 2005-08-15; First posted 2005-08-17 (Estimated); Last update posted 2008-09-22 (Estimated); Status verified 2008-09

CONDITIONS: Psoriasis
Keywords: Previously enrolled on a MEDI-507 for psoriasis
MeSH Terms: conditions — Psoriasis | interventions — siplizumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

INTERVENTIONS:
Other: Follow up from previous treatment with MEDI-507 — There will be no investigational drugs administered under this protocol.

SUMMARY:
The purpose of this study is to evaluate the long-term safety and profile of psoriasis patients who have completed participation in a previous study and who received treatment with MEDI-507.

DETAILED DESCRIPTION:
This study will evaluate the long-term safety and lymphocyte repletion profile of psoriasis patients who have completed participation in a previous study and who received treatment with MEDI-507. Patients must have had an ALC > 30% lower than baseline (defined as baseline prior to any MEDI-507 exposure); or an absolute CD4 count of < 250 cells/uL. This study will also evaluate the development and durability of anti-MEDI-507 antibodies.

ELIGIBILITY:
Inclusion Criteria:

* The patient has previously completed participation (i.e., completed per protocol, including any long term follow-up; or discontinued from the study due to withdrawal of consent, loss to follow-up, or other reason) in a Medimmune, Inc. study of MEDI-507 in psoriasis in which they received MEDI-507 (or placebo for patients who participated in a blinded placebo-controlled study of MEDI-507, and for whom the treatment assignment in that study has not been unblinded at the time of entry into this study)
* The patient had an absolute lymphocyte count (ALC) > 30% lower than baseline (defined as baseline prior to any MEDI-507 exposure; or, for patients whose treatment assignments have not been unblinded at the time of entry into this study, drug exposure) at his/her final visit (excluding any long-term follow-up visits) in the most recent Medimmune, Inc. study in which the patient participated; or the patient had an absolute CD4 count of < 250 cells/uL at his/her final visit (including any protocol-specific long-term follow up) in the most recent Medimmune, Inc. study in which the patient participated.
* Written informed consent obtained from the patient

Exclusion Criteria:

* There are no exclusion criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient has previously completed participation
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2002-08; Primary Completion 2003-10 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara White, M.D., Study Director — MedImmune LLC
Locations (21):
- United States (7):
  - Dermatology Research Clinic, Little Rock, Arkansas
  - Cherry Creek Dermatology, Denver, Colorado
  - Atlanta Dermatology, Vein & Research Center, LLC, Alpharetta, Georgia
  - Future Care Studies, Springfield, Massachusetts
  - Washington University, Dermatology Clinical Trials Unit, St Louis, Missouri
  - VA Medical Center, Nashville, Tennessee
  - Northwest Kinetics, Tacoma, Washington
- Belgium (2):
  - Universitaur Ziekenhuis Gent, Ghent
  - CHU Centre Ville, Liège
- Canada (3):
  - Capital District Health Authority, QE II Health Sciences Center, Halifax, Nova Scotia
  - International Dermatology Research, Montreal, Quebec
  - Innovaderm Research, Montreal
- France (3):
  - Hotel Dieu/Clinque Dermatologique, Nantes
  - Hospital Saint-Louis Service de Dermatologie 1, Paris
  - Hospital Haut Leveque CHU Sud -Service de Dermatologie, Pessac
- Germany (5):
  - Universitataskilinkum der TU Dresden, Dresden
  - Universitatsklinikum Hautklinik, Düsseldorf
  - Klinikum de Johann - Wolfgang Goethe Universitate Frankfurt, Frankfurt
  - St. Urban, Dermatologie, Freiburg im Breisgau
  - Universitatsklinikum Hautklinik, Tübingen
- Academisch Medisch Centrum/Universiteit van Amsterdam (AMC/UvA), Amsterdam, Netherlands